CLINICAL TRIAL: NCT02123888
Title: Simultaneous Cone Beam Computed Tomography (CBCT) Acquisition During Arc Radiotherapy
Brief Title: Simultaneous CBCT Acquisition During Arc Radiotherapy
Acronym: SCART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sally Falk (Other)
Responsible Party: Sponsor-Investigator, Sally Falk, Clinical Trial Project Manager, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10_RADIO_94
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Prostate Cancer; Lung Cancer
Keywords: Prostate; Lung
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cone Beam Computed Tomography (Experimental): Simultaneous Cone Beam Computed Tomography acquisition during arc radiotherapy.
  Interventions: Radiation: Cone Beam Computed Tomography

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography — Simultaneous Cone Beam Computed Tomography acquisition during arc radiotherapy

SUMMARY:
The cone beam image is a part of the radiotherapy treatment machine and uses lower energy xrays as the head of the radiotherapy machine moves around the patient in a circle. This takes pictures that give 3-dimensional information, somewhat like a CT scan. These images are better at showing the position of the tumour and surrounding soft tissues than the standard xrays that were previously used. Cone Beam Imaging Technology is not new and has been used regularly at The Christie for many years. The standard cone beam scan is taken before the actual radiotherapy treatment or after the treatment has been delivered.

Volumetric Modulated Arc Therapy (VMAT or Arc Radiotherapy) is a novel method of delivering radiotherapy that involves the continuous movement of the radiotherapy treatment machine head around the patient and MLC during radiation. Arc radiotherapy has been clinically implemented at The Christie for prostate radiotherapy treatments and work is in progress for implementation in lung radiotherapy. The continuous gantry rotation inherent to VMAT delivery makes this simultaneous imaging possible, although there are concerns associated with the impact that this may have on patient dose and image quality.

The aim of this research is to assess whether the image quality of cone beam scans taken during treatment are as good as standard cone beam scans taken before or after treatment used to determine the accuracy of patient position and the tumour coverage by radiotherapy.

ELIGIBILITY:
Inclusion Criteria for prostate cancer patients:

* Patients to be treated with radical RT for prostate cancer
* Patients to be treated with VMAT
* ECOG performance status 0-2
* Patients must be able to receive and understand verbal and written information regarding the study and give written, informed consent

Inclusion Criteria for lung cancer patients:

* A histological or cytological diagnosis of non-small cell lung cancer or small cell lung cancer
* Patients to be treated with radical RT or SBRT
* Patients to be treated with VMAT
* ECOG performance status 0-2
* Patients must be able to receive and understand verbal and written information regarding the study and give written, informed consent
* Female patients must meet one of the following criteria - postmenopausal for a minimum of one year, surgically sterile, not pregnant, confirmed by β-HCG blood test and willing to use adequate contraception during study participation, not breastfeeding

Exclusion Criteria for prostate cancer patients:

* Clinical judgement by the investigator that the patient should not participate in the study
* Patients in clinical trials of new investigational medicinal products or treatment regimens unless there is written, prior agreement that the patient can also consent to this study, and that clinical data can also be used for this study
* Prior radiotherapy or surgery in the pelvis that can make identification of normal anatomy difficult

Exclusion criteria for lung cancer patients:

* Clinical judgement by the investigator that the patient should not participate in the study
* Patients in clinical trials of new investigational medicinal products or treatment regimens unless there is written, prior agreement that the patient can also consent to this study, and that clinical data can also be used for this study
* Prior radiotherapy or surgery in the region of interest that can make identification of normal anatomy difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Equivalence of image quality | 12 months
  To show equivalence of image quality from simultaneous CBCT acquisition during delivery of arc radiotherapy with that obtained from conventional CBCT acquisition in lung and prostate patients, as assessed by user-questionnaires.

SECONDARY OUTCOMES:
Quantify inter-observer variation | 12 months
  To quantify inter-observer variation in interpretation of anatomy, as assessed by questionaires.
Quantify inter-observer variation | 12 months
  To quantify inter-observer variation in delineation of specific structures on CBCT scans.
Quantify impact on treatment times. | 12 months
  To quantify the impact of simultaneous CBCT scans on treatment times.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, MD PhD, Principal Investigator — The Christie NHS Foundation Trust; Ananya Choudhury, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom